CLINICAL TRIAL: NCT01102660
Title: A Randomized, Double-Blind, Double-Dummy, Placebo And Active Controlled Two Period Four Treatment Cross-Over Clinical Trial To Examine The Pain Relief Of PH-797804 Alone Or With Naproxen In Subjects With Flare-Enriched Osteoarthritis Of The Knee
Brief Title: Clinical Trial to Examine the Pain Relief of PH-797804 Alone Or With Naproxen in Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A6631026
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Osteoarthritis
Keywords: Knee osteoarthritis; clinical trial; cross-over
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — PH 797804; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment Sequence 1 (Other)
  Interventions: Drug: PH-797804; Drug: Placebo
- Treatment Sequence 2 (Other)
  Interventions: Drug: Placebo; Drug: PH-797804
- Treatment Sequence 3 (Other)
  Interventions: Drug: Naproxen; Drug: Naproxen + PH-797804
- Treatment Sequence 4 (Other)
  Interventions: Drug: Naproxen + PH-797804; Drug: Naproxen

INTERVENTIONS:
Drug: PH-797804 — Tablet, 6 mg once daily for 2 weeks
  Arms: Treatment Sequence 1
Drug: Placebo — Tablet, 0 mg once daily for 2 weeks
  Arms: Treatment Sequence 1
Drug: Placebo — Tablet, 0 mg once daily for 2 weeks
  Arms: Treatment Sequence 2
Drug: PH-797804 — Tablet, 6 mg once daily for 2 weeks
  Arms: Treatment Sequence 2
Drug: Naproxen — Tablet, 500 mg twice daily for 2 weeks
  Arms: Treatment Sequence 3
Drug: Naproxen + PH-797804 — Tablet, 500 mg twice daily for 2 weeks and Tablet, 6 mg once daily for 2 weeks
  Arms: Treatment Sequence 3
Drug: Naproxen + PH-797804 — Tablet, 500 mg twice daily for 2 weeks and Tablet, 6 mg once daily for 2 weeks
  Arms: Treatment Sequence 4
Drug: Naproxen — Tablet, 500 mg twice daily for 2 weeks
  Arms: Treatment Sequence 4

SUMMARY:
PH-797804 is a potent inhibitor of inflammatory mediators that have a potential role in pain signalling following nerve injury and inflammation. Blocking such mediators may potentially have a therapeutic benefit by reducing pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including, the ages of 18 and 75 years. Females must be of non-childbearing potential.
* Diagnosis of osteoarthritis of the knee based on American College of Rheumatology criteria with X-ray confirmation (a Kellgren-Lawrence X-ray grade of ≥2.

Exclusion Criteria:

* History of diseases other than osteoarthritis that may involve the index knee.
* Other severe pain that impairs the assessment of osteoarthritis of pain.
* Electrocardiogram abnormalities.
* History of gastrointestinal disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Western Ontario & McMaster Osteoarthritis Index Pain Score | 2 weeks

SECONDARY OUTCOMES:
Western Ontario & McMaster Osteoarthritis Index Stiffness Score | 2 weeks
Western Ontario & McMaster Osteoarthritis Index Physical Function Score | 2 weeks
Western Ontario & McMaster Osteoarthritis Index Total Score | 2 weeks
Daily Pain Rating Scale | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (23):
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Spring Valley, California
  - Pfizer Investigational Site, Valley Village, California
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, Hyannis, Massachusetts
  - Pfizer Investigational Site, New Bedford, Massachusetts
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Wilmington, North Carolina
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Pawtucket, Rhode Island
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631026&StudyName=Clinical%20Trial%20to%20Examine%20the%20Pain%20Relief%20of%20PH-797804%20Alone%20Or%20with%20Naproxen%20in%20Subjects%20with%20Osteoarthritis%20of%20the%20Knee